CLINICAL TRIAL: NCT05054569
Title: Developing and Pre-Testing an eHealth Group Intervention for Young Adult Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Principal Investigator, Rina Fox, Research Assistant Professor, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: NU 20CC18; IRG-18-163-24 (Other Grant/Funding Number: American Cancer Society); STU00214055 (Other: Northwestern University Institutional Review Board)
Record Dates: First submitted 2021-09-03; First posted 2021-09-23 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2021-12

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 10-week eHealth intervention (Experimental): Weekly video conference groups led by a trained facilitator
  Interventions: Behavioral: Cognitive-Behavioral Stress Management and Health Education

INTERVENTIONS:
Behavioral: Cognitive-Behavioral Stress Management and Health Education — Participants will attend group sessions with a trained facilitator held over videoconference. Sessions will each last 2 hours and will be held once weekly for 10 weeks. Sessions will include Cognitive-Behavioral Stress Management and health education content.

SUMMARY:
The purpose of this study is to develop and pre-test an eHealth group intervention for young adult cancer survivors.

DETAILED DESCRIPTION:
In the first part of this study, the investigators adapted an evidence-based intervention for improving HRQOL to better meet the needs of young adult cancer survivors, and then conducted focus groups with young adult cancer survivors to get feedback on the adapted intervention. In the second part of the study, the investigators will conduct a single-arm pilot trial in which the adapted intervention will be delivered over videoconference via weekly group meetings with a trained facilitator over the course of 10 weeks.

ELIGIBILITY:
Inclusion Criteria:

* age 18-39 years at the time of participation
* diagnosed with a non-metastatic primary cancer between 18-39 years old
* completed primary cancer treatment (excepting hormone therapy) 1 month to 5 years prior to enrollment
* able to speak and read English
* access to internet or cellular connectivity with sufficient bandwidth to participate in videoconferences

Exclusion Criteria:

* metastatic disease
* psychiatric or neurological disorders that could interfere with study participation
* considered part of a vulnerable population

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2021-12-15 (Actual)

PRIMARY OUTCOMES:
Acceptability of the adapted intervention | Over the course of the 10-week intervention, beginning with the first weekly session through the tenth weekly session
  Participants will report their satisfaction with individual sessions through brief weekly surveys.
Acceptability of the adapted intervention | Over the course of the 10-week intervention, beginning with the first weekly session through the tenth weekly session
  The number of sessions attended, out of a maximum of 10, will be tracked.
Acceptability of the adapted intervention | Immediately after the intervention
  Immediately after the intervention participants will report their satisfaction with the full program through a brief survey.

SECONDARY OUTCOMES:
Change in health-related quality of life (HRQOL) from baseline to immediately after the intervention | Baseline and immediately after the intervention
  Participants will complete the 27-item Functional Assessment of Cancer Therapy - General. Scores range from 0 to 108, with higher scores reflecting better quality of life.
Change in symptom burden from baseline to immediately after the intervention | Baseline and immediately after the intervention
  Participants will complete a modified version of the Edmonton Symptom Assessment Scale, which assesses 10 common cancer-related symptoms each on a numerical rating scale ranging from 0 to 10. Higher scores indicate greater symptom burden.
Change in cancer-related distress from baseline to immediately after the intervention | Baseline and immediately after the intervention
  Participants will complete the 22-item Impact of Event Scale-Revised. Scores range from 0 to 88, with higher scores indicating greater cancer-related distress.
Change in stress management skills self-efficacy from baseline to immediately after the intervention | Baseline and immediately after the intervention
  Participants will complete subscales from the Measure of Current Status. Subscale scores range from 0 to 8, 0 to 12, or 0 to 20 depending on the subscale. Higher scores indicate more of the construct being assessed.
Change in coping from baseline to immediately after the intervention | Baseline and immediately after the intervention
  Participants will complete the Brief Coping Orientation to Problems Experienced scale, which yields 14 two-item subscales. Subscale scores range from 2 to 8, with higher scores indicating greater usage of the coping strategy being assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern University Feinberg School of Medicine, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fox RS, Badger TA, Moya S, Gudenkauf LM, Nelson MA, O'Neill RM, Leete JJ, Friedman SE, Katsanis E, Victorson DE, Sanford SD, Penedo FJ, Antoni MH, Oswald LB. An HRQOL Proof-Of-Concept Analysis of the eHealth TOGETHER Intervention for Adolescent and Young Adult Cancer Survivors: A Brief Report. Psychooncology. 2025 Jul;34(7):e70234. doi: 10.1002/pon.70234. PMID 40879639
- [Derived] Oswald LB, Lyleroehr M, Gudenkauf LM, Armstrong GE, Tometich DB, Sanford SD, Loecher N, Geiss C, Rodriguez Y, Scheel KL, Nieves-Lopez A, Jim HSL, Gonzalez BD, Antoni MH, Penedo FJ, Reed D, Katsanis E, Salsman JM, Victorson D, Fox RS. Development and initial testing of TOGETHER-YA: an eHealth-delivered and group-based psychosocial intervention for young adult cancer survivors. Support Care Cancer. 2022 Dec;30(12):10067-10076. doi: 10.1007/s00520-022-07382-y. Epub 2022 Oct 14. PMID 36229547